CLINICAL TRIAL: NCT05916157
Title: A Post-marketing Observational Study for ABBV-951 in Patients Diagnosed With Advanced Parkinson's Disease (aPD)
Brief Title: An Observational Study of Subcutaneous Infusion of ABBV-951 to Assess Change in Disease Activity and Adverse Events In Adult Japanese Participants With Advanced Parkinson's Disease
Status: Recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P23-529
Record Dates: First submitted 2023-06-15; First posted 2023-06-23 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Parkinson's Disease (PD)
Keywords: Parkinson's Disease (PD); advanced Parkinson's disease (aPD); ABBV-951
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ABBV-951: Participants will receive ABBV-951 as prescribed by their physician.

SUMMARY:
Parkinson's disease (PD) is a neurological condition, which affects the brain. Some symptoms of PD are tremors, stiffness, and slowness of movement. The purpose of this study is to assess how safe and effective ABBV-951 is in treating participants with Parkinson's disease in real world setting.

ABBV-951 is an approved drug being developed for the treatment of PD in Japan. Approximately 250 adult participants over 15 years with a diagnosis of PD who are prescribed ABBV-951 by their physicians will be enrolled in this study across Japan.

Participants will receive ABBV-951 as prescribed their physician and followed for 52 weeks.

There is expected to be no additional burden for participants in this trial. Study visits may be conducted on-site or virtually as per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with advanced Parkinson's disease (aPD).
* Prescribed ABBV-951 as physicians' decision according to the approved label for treatment of aPD.
* Given informed consent (or by her/his legal representative, if it's a requirement from the participating hospital/clinic) for participating this study.

Exclusion Criteria:

* Prior treatment with ABBV-951 for PD.
* Currently participating in interventional clinical trials.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult participants who are prescribed ABBV-951 for the treatment of advanced Parkinson's disease (aPD).
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing Infusion Site Infections | Up to 52 Weeks
  Percentage of participants with infusion site infections following the commencement of ABBV-951 will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (16):
- Japan (16):
  - Saiseikai Matsuyama Hospital /ID# 276259, Matsuyama, Ehime
  - National Hospital Organization Asahikawa Medical Center /ID# 269115, Asahikawa, Hokkaido
  - Ryugasaki Saiseikai Hospital /ID# 264435, Ryūgasaki, Ibaraki
  - University of Tsukuba Hospital /ID# 268353, Tsukuba, Ibaraki
  - Okatsu Hospital /ID# 262781, Kagoshima, Kagoshima-ken
  - University Hospital Kyoto Prefectural University of Medicine /ID# 267445, Kyoto, Kyoto
  - Sendai Nishitaga National Hospital /ID# 268349, Sendai, Miyagi
  - Fujimoto General Hospital /ID# 277287, Miyakonojo-shi, Miyazaki
  - Shiga University of Medical Science Hospital /ID# 265637, Ōtsu, Shiga
  - Dokkyo Medical University Hospital /ID# 269116, Mibu, Tochigi
  - Juntendo University Hospital /ID# 264438, Bunkyo-ku, Tokyo
  - Nitobe Memorial Nakano General Hospital /ID# 275668, Nakano-ku, Tokyo
  - National Center of Neurology and Psychiatry - Kodaira /ID# 267372, Xiaoping City, Tokyo
  - National Hospital Organization Utano Hospital /ID# 268350, Kyoto
  - Okayama Neurology Clinic /ID# 269117, Okayama
  - Municipal Toyonaka Hospital /ID# 271277, Toyonaka

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P23-529